CLINICAL TRIAL: NCT01590342
Title: Efficacy of Diclofenac for Patients With Acute Submassive Pulmonary Embolism: a Randomized Clinical Trial
Brief Title: Diclofenac for Submassive PE
Acronym: AINEP-1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, David Jimenez, Clinical researcher, Ministry of Health, Spain
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-000247-27
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Right ventricular dysfunction; Prognosis; Inflammation
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right; Inflammation | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — Diclofenac 75 mg, two doses
  Arms: Diclofenac
Drug: Placebo — Placebo, two doses
  Arms: Placebo

SUMMARY:
The primary objective is to demonstrate the clinical benefits of diclofenac (added to standard anticoagulant therapy) over placebo in normotensive patients with acute symptomatic pulmonary embolism and right ventricular dysfunction.

The secondary objective is to assess the safety after administration of diclofenac in normotensive patients with acute symptomatic pulmonary embolism and right ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic PE confirmed by multidetector CT angiography, a high-probability V/Q scan, or by the presence of deep vein thrombosis confirmed by lower limb ultrasound testing in patients with nonconclusive V/Q scan;
2. first symptoms occurring ten days or less before randomization;
3. haemodynamic stability (systolic blood pressure > 100 mm Hg, no need of inotropic support, pulmonary resuscitation, intubation or thrombolytic treatment);
4. right ventricular dysfunction assessed by transthoracic echocardiography within the first 12 hours after diagnosis of PE;
5. signed informed consent.

Exclusion Criteria:

1. Previous diagnosis of chronic thromboembolic pulmonary hypertension;
2. active bleeding, or clinically relevant bleeding in the previous month before diagnosis of PE;
3. peptic ulcer;
4. major surgery, or severe trauma in the previous month before diagnosis of PE;
5. indication for chronic anticoagulation;
6. pregnancy or breast feeding;
7. renal insufficiency (serum creatinine > 2 mg/dL) or severe hepatic impairment;
8. hypersensitivity to diclofenac, sodium metabisulfite, or acetylsalicylic acid;
9. bronchial asthma;
10. severe congestive heart failure;
11. inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Right ventricular dysfunction assessed by transthoracic echocardiography | 36-48 hours after administration of the first dose of diclofenac/placebo

SECONDARY OUTCOMES:
Right ventricular dysfunction assessed by transthoracic echocardiography | Seven days after administration of diclofenac/placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Jimenez, MD, PhD, Study Chair — Ramon y Cajal Hospital, IRYCIS
Locations (1):
- Ramon y Cajal Hospital, IRYCIS, Madrid, Spain

REFERENCES:
- [Derived] Jimenez D, Nieto R, Corres J, Fernandez-Golfin C, Barrios D, Morillo R, Quezada CA, Huisman M, Yusen RD, Kline J. Diclofenac for reversal of right ventricular dysfunction in acute normotensive pulmonary embolism: A pilot study. Thromb Res. 2018 Feb;162:1-6. doi: 10.1016/j.thromres.2017.12.002. Epub 2017 Dec 5. PMID 29247809